CLINICAL TRIAL: NCT04195126
Title: Early Haemadsorption Treatment of Major Burn Trauma Patients
Brief Title: Early Haemadsorption in Major Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7066 - PTE 2018
Record Dates: First submitted 2018-05-05; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Burns; Multiple Organ Failure; Shock; Organ Dysfunction Syndrome, Multiple; Renal Dysfunction; Cytokine Storm
MeSH Terms: conditions — Burns; Multiple Organ Failure; Shock; Renal Insufficiency; Cytokine Release Syndrome

STUDY DESIGN:
Intervention Model Description: Patients included in our study are randomised into treatment or control groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors are unaware of the patient groups. Treated patients are not informed regarding randomisation results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients are treated according to most recent guidelines in burn trauma and corresponding emergency and intensive therapy. All patients included are treated with early continous veno-venal renal replacement therapy.
- Treatment group (Active Comparator): Besides treatment strategies of the control group, the investigators start early haemadsorption treatment right after patient admission (and inclusion).
  Interventions: Device: CytoSorb haemadsorption device

INTERVENTIONS:
Device: CytoSorb haemadsorption device — CytoSorb (Cytosorbents Inc.) aspecific blood purification device used in an extracorporeal circulation system without dialysis column. Anticoagulation is managed by siodium citrate-Calcium system, using the Gambro CVVHDF capable device.
  Arms: Treatment group

SUMMARY:
Major deep burns (>20% body surface, involving deep skin layers) and associated severe inflammatory reaction and their complication are one of the biggest challenge of intensive care. Haemoadsorption therapy, including the CytoSorb treatment is a promising novel therapeutic approach, but only case-studies are available in the literature yet. Based on data from septic shock patient treatment the investigators hypothesize that CytoSorb is beneficial in early treatment of burns. The investigators aim to conduct a randomised-controlled study to assess the clinical effectiveness (based on score systems including MODS, SOFA, APACHE II, KDIGO, ABSI), 7 and 28 days survival, intensive care length of stay, length of mechanical ventilation, resuscitation fluid need and ino/vasopressor drug doses and the presence and severity of organ dysfunctions, particularly renal dysfunction. The investigatora plan to conduct basic research to elucidate the pathophysiological background of clinical effect, including the measurement of inflammatory and anti-inflammatory cytokines, presence and severity of oxidative stress (lipid peroxidation, protein oxidation, reduced/oxidised glutathion levels) and organ dysfunction markers (kidney injury molecule -1, neutrophil gelatinase-associated lipocalin, cystatin-C, uromodulin).

ELIGIBILITY:
Inclusion Criteria:

* informed consent of our patient or next of kin,
* TBSA >20% with 2/b depth of burn

Exclusion Criteria:

* non-thermal burn injury,
* need for acute haemodialysis (intoxication),
* immunosuppressive treatment, chronic steroid use (> 3 months),
* known malignant disease,
* end-stage renal insufficiency or renal transplantation,
* Child C hepatic cirrhosis,
* gravidity,
* potentially lethal burn (Baux index >120) or comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
7 days mortality | Survival rate is assessed in the 7th admission day.
  The investigators assess the intensive care and post-intensive care mortality of our patients.
28 days mortality | Survival rate is assessed in the 28th admission day.
  The investigators assess the intensive care and post-intensive care mortality of our patients.

SECONDARY OUTCOMES:
Levels of inflammatory and anti-inflammatory cytokines during treatment | Samples are gathered on inclusion and 8, 16, 24, 48, 72, 96, 120, 148, 168 hours following. Measured data points are selected by screening. All measurements are carried out in one lot. Data will be presented in arbitrary units.
  The investigators assess the course of pro- and anti-inflammatory cytokines during ICU stay for both patient groups. Cytokines are screened by the Human Cytokine Array. Selected markers are measured individually.
Markers of oxidative stress (ROS production, MDA levels, tyrosine isomers) | Samples are gathered on inclusion and 8, 16, 24, 48, 72, 96, 120, 148, 168 hours following. Measured data points are selected by screening. All measurements are carried out in one lot.
  The investigators follow the severity of oxidative stress in both groups.
Intensive Care Unit length of stay | Length of intensive care for each patient (days), data is registered through ICU discharge of the patient, an average of 1 month.
  The investigators assessed the duration of ICU stay (in days)
Volume resuscitation fluid need of our patients. | Results are summarised daily for our patients during the first week following inclusion.
  The investigators assess the primary volume resuscitation need of our patients.
Vasopressor need of our patients. | Results are summarised daily for our patients during the first week following inclusion.
  The investigators assess the daily average vasopressor dose of our patients.
Length of mechanical ventilation (if needed). | Length of mechanical ventillation (days). Data is registered through patient discharge from ICU, an average of 1 month.
  The investigators assess whether CytoSorb treatment reduce the length of mechanical ventilation
Severity of organ failures according to SOFA point system | Assessed daily for each patient during the first week of our study. Worst results are registered.
  The investigators assess the severity of multiple organ dysfunction/failure according to SOFA score.

CONTACTS AND LOCATIONS:
Overall Officials: Gábor Woth, MD PhD, Principal Investigator — University of Pécs, Dept. of Anaesthesia and Intensive Care
Locations (1):
- University of Pécs, Dept. of Anaesthesia and Intensive Care, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: Undecided
The investigators plan to share patient clinical data and laboratory measurement results following study result publication.